CLINICAL TRIAL: NCT01086657
Title: VRC 310: An Open-Label, Randomized Ph I: Healthy Adults of Prime-Boost Intervals w/Monovalent Influenza Virion (H5N1) Vaccine, A/Indonesia/05/2005 (Sanofi Pasteur, Inc), Administered Alone or Following Recombinant H5 DNA Vaccine
Brief Title: An Open-Label, Randomized Phase I Study in Healthy Adults of the Safety and Immunogenicity of Prime-Boost Intervals With Monovalent Influenza Subunit Virion (H5N1) Vaccine, A/Indonesia/05/2005 (Sanofi Pasteur, Inc.) Administered Alone or Following Re...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100069; 10-I-0069
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-12

CONDITIONS: Influenza A Virus, H5N1 Subtype
Keywords: Bird Flu; Avian Influenza; Healthy; Immunity; Prevention; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza in Birds | interventions — Vaccines

ARMS (6):
- Group 1 (Experimental): Inactivated H5N1 Vaccine at Enrollment and inactivated H5N1 Vaccine at Week 24
  Interventions: Biological: VRC-AVIDNA036-00-VP; Biological: Monovalent Influenza Subunit Virion (Inactive H5N1) Vaccine
- Group 2 (Experimental): H5 DNA Vaccine at Enrollment and Inactivated H5N1 Vaccine at Week 4
  Interventions: Biological: VRC-AVIDNA036-00-VP
- Group 3 (Experimental): H5 DNA Vaccine at Enrollment and Inactivated H5N1 Vaccine at Week 8
  Interventions: Biological: VRC-AVIDNA036-00-VP
- Group 4 (Experimental): H5 DNA Vaccine at Enrollment and Inactivated H5N1 Vaccine at Week 12
  Interventions: Biological: VRC-AVIDNA036-00-VP
- Group 5 (Experimental): H5 DNA Vaccine at Enrollment and Inactivated H5N1 Vaccine at Week 16
  Interventions: Biological: VRC-AVIDNA036-00-VP
- Group 6 (Experimental): H5 DNA Vaccine at Enrollment and Inactivated H5N1 Vaccine at Week 24
  Interventions: Biological: VRC-AVIDNA036-00-VP

INTERVENTIONS:
Biological: VRC-AVIDNA036-00-VP — H5 DNA Vaccine
Biological: Monovalent Influenza Subunit Virion (Inactive H5N1) Vaccine — Inactive H5N1 Vaccine
  Arms: Group 1

SUMMARY:
Background:

- New vaccines against avian influenza, also known as "bird flu," are being developed and require testing to determine if they are safe and effective and whether they have any side effects. Researchers are interested in testing two experimental avian influenza vaccines to see whether they are safe, if there are any side effects from the vaccines, and how the body's immune response differs in response to different vaccination schedules. One vaccine is an inactivated vaccine (made with killed or weakened influenza) and one is a DNA vaccine that allows the body to use vaccine to make an immune system response to a specific part of an avian influenza protein.

Objectives:

* To determine the safety and potential side effects of two experimental vaccines against avian influenza.
* To evaluate whether the time between the two experimental vaccine injections affects the immune response to the vaccine.

Eligibility:

- Healthy individuals between 18 and 60 years of age.

Design:

* Participants will be randomly divided (by chance) into six groups to receive two injections of vaccine at different intervals. One group will receive only the inactivated vaccine, while the other groups will receive the DNA vaccine followed by the inactivated vaccine at different intervals (e.g., 4 weeks, 8 weeks, 12 weeks, 16 weeks or 24 weeks later).
* Participants will remain at the clinical center for at least 30 minutes after each vaccination. A few days after each injection, participants will contact staff by telephone or have a clinic visit. Participants will also be asked to complete a diary card at home for 5 days to keep track of temperature changes, injection site skin changes, and other effects.
* Four weeks after the first injection, participants will return for a clinic visit and to provide blood samples for testing.
* Two weeks after the second injection, participants will return for a clinic visit and provide blood samples (collected through apheresis) to provide information on immune response to the vaccine.

DETAILED DESCRIPTION:
An Open-Label, Randomized Phase I Study in Healthy Adults of the Safety and Immunogenicity of Prime-Boost Intervals with Monovalent Influenza Subunit Virion (H5N1) Vaccine, A/Indonesia/05/2005 (Sanofi Pasteur, Inc), Administered Alone or Following Recombinant DNA Plasmid (H5) Vaccine, VRC-AVIDNA036-00-VP (VRC, NIAID)

Study Design:

This is a Phase I, randomized, open-label study to evaluate the safety, tolerability, and immunogenicity of prime-boost vaccination regimens against the influenza virus hemagglutinin H5. One group will receive A/Indonesia/05/2005 (inactivated H5N1) vaccine as both prime and boost, and the other groups will receive the VRC-AVIDNA036-00-VP (DNA) vaccine as prime with inactivated H5N1 boost but with various boost intervals. The VRC 310 study will provide data from different prime-boost schedules to identify whether homologous or heterologous schedules result in a better antibody response as well as which interval of time between vaccinations is associated with the best immune response. The hypothesis is that all of the study regimens will be safe for human administration and will elicit antibody and T cell responses against the H5 protein. The primary objectives are to evaluate the safety and tolerability of the investigational vaccine regimens, at a dose of 4 mg for the DNA vaccine and 90 microg for the inactivated H5N1, in healthy adults. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine regimens and identification of an interval between prime and boost that has the highest frequency of strong immune responses.

Product Description:

The inactivated H5N1 vaccine is monovalent subunit virion vaccine, A/Indonesia/05/2005 clade 2, manufactured by Sanofi Pasteur, Inc (Swiftwater, PA). Vaccine vials will be supplied at 90 microg/0.5mL. The VRC-AVIDNA036-00-VP vaccine was developed and manufactured by VRC, NIAID and is composed of a single closed-circular DNA plasmid that encodes the H5 protein with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each vaccination will be administered intramuscularly (IM) in the deltoid muscle using needle and syringe for the H5N1 vaccine and the Biojector 2000 Needle-Free Injection Management System (Biojector) for the DNA vaccine.

Subjects:

A total of 60 healthy adults, ages 18-60 years will be enrolled.

Study Plan:

Subjects will be simultaneously randomized equally into one of 6 groups. Subjects and clinicians will be blinded to group assignment until Day 0 following completion of the enrollment. At the point of enrollment the randomly assigned regimen will become known to subjects and clinicians. Subjects will receive two injections on the schedule shown in the schema. The protocol requires 5 or 6 clinic visits, depending upon the group, and telephone follow-up contact after the first study injection and 24 weeks after the second study injection. Additional optional visits may be conducted at study weeks 48 and 72 to collect blood for evaluation of immune response durability.

Study Duration:

Each participant will complete clinical follow up through 24 weeks after the second vaccination. Duration of the expected time on study will vary from 28 to 48 weeks depending upon the Group, but may be extended to 72 weeks after enrollment for subjects who agree to complete the optional research blood drawas.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

18 to 60 years old.

Available for clinical follow-up for up to 32 weeks after enrollment.

Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.

Complete an Assessment of Understanding (AoU) questionnaire prior to enrollment and verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to donate blood for sample storage to be used for future research.

In good general health without clinically significant medical history.

Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) < 40 within the 56 days prior to enrollment.

Laboratory Criteria within 56 days prior to enrollment:

Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to13.5 g/dL for men

White blood cells (WBC) = 3,300-12,000 cells/mm(3)

Differential either within institutional normal range or accompanied by site physician approval

Total lymphocyte count greater than or equal to 800 cells/mm3

Platelets = 125,000 - 500,000/mm(3)

Alanine aminotransferase (ALT) < 1.25 x upper limit of normal (ULN)

Serum creatinine less than or equal to 1 x ULN (less than or equal to1.3 mg/dL for females; less than or equal to1.4 mg/dL for males)

Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]

Women Specific:

Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential.

A female subject must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Agrees to be heterosexually inactive at least 21 days prior to enrollment and through8 weeks after last injection,

OR

Agrees to consistently practice contraception at least 21 days prior to enrollment and through 8 weeks after last injection by one of the following methods:

* condoms, male or female, with or without a spermicide;
* diaphragm or cervical cap with spermicide;
* intrauterine device;
* contraceptive pills, patch, implant or any other FDA-approved contraceptive method;
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply.

Women Specific:

Breast-feeding or planning to become pregnant during the first 28 weeks after enrollment in the study.

Subject has received any of the following substances:

Systemic immunosuppressive medications or cytotoxic medications within the 12 weeks prior to enrollment. [With the exception that a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]

Blood products within 112 days (16 weeks) prior to HIV screening

Immunoglobulin within 56 days (8 weeks) prior to HIV screening

Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration

Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days (2 weeks) of initial study vaccine administration

Current anti-TB prophylaxis or therapy

Previous H5 avian influenza investigational vaccine.

Subject has a history of any of the following clinically significant conditions:

Contraindication to receiving an FDA approved current seasonal influenza vaccination (e.g., egg allergy)

Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.

Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

Thyroid disease that is not well controlled.

Idiopathic urticaria within the past year

Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.

Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.

Allergic reaction to aminoglycoside antibiotics.

Guillain-Barr Syndrome.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02-25; Primary Completion 2011-12-12 (Actual); Study Completion 2011-12-12 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events, including clinical, laboratory and local and systemic reactogenicity

SECONDARY OUTCOMES:
Immunogenicity as measured by humoral and cellular assays.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Taubenberger JK, Reid AH, Lourens RM, Wang R, Jin G, Fanning TG. Characterization of the 1918 influenza virus polymerase genes. Nature. 2005 Oct 6;437(7060):889-93. doi: 10.1038/nature04230. PMID 16208372
- [Derived] Andrews SF, Raab JE, Gorman J, Gillespie RA, Cheung CSF, Rawi R, Cominsky LY, Boyington JC, Creanga A, Shen CH, Harris DR, Olia AS, Nazzari AF, Zhou T, Houser KV, Chen GL, Mascola JR, Graham BS, Kanekiyo M, Ledgerwood JE, Kwong PD, McDermott AB. A single residue in influenza virus H2 hemagglutinin enhances the breadth of the B cell response elicited by H2 vaccination. Nat Med. 2022 Feb;28(2):373-382. doi: 10.1038/s41591-021-01636-8. Epub 2022 Feb 3. PMID 35115707
- [Derived] Ledgerwood JE, Zephir K, Hu Z, Wei CJ, Chang L, Enama ME, Hendel CS, Sitar S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 310 Study Team. Prime-boost interval matters: a randomized phase 1 study to identify the minimum interval necessary to observe the H5 DNA influenza vaccine priming effect. J Infect Dis. 2013 Aug 1;208(3):418-22. doi: 10.1093/infdis/jit180. Epub 2013 Apr 30. PMID 23633407
- [Derived] Khurana S, Wu J, Dimitrova M, King LR, Manischewitz J, Graham BS, Ledgerwood JE, Golding H. DNA priming prior to inactivated influenza A(H5N1) vaccination expands the antibody epitope repertoire and increases affinity maturation in a boost-interval-dependent manner in adults. J Infect Dis. 2013 Aug 1;208(3):413-7. doi: 10.1093/infdis/jit178. Epub 2013 Apr 30. PMID 23633404
- [Derived] Ledgerwood JE, Wei CJ, Hu Z, Gordon IJ, Enama ME, Hendel CS, McTamney PM, Pearce MB, Yassine HM, Boyington JC, Bailer R, Tumpey TM, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 306 Study Team. DNA priming and influenza vaccine immunogenicity: two phase 1 open label randomised clinical trials. Lancet Infect Dis. 2011 Dec;11(12):916-24. doi: 10.1016/S1473-3099(11)70240-7. Epub 2011 Oct 3. PMID 21975270